CLINICAL TRIAL: NCT02198768
Title: Functional Outcome After Ankle Fractures and Ankle Fracture-Dislocations: A Prospective Study
Brief Title: Ankle Fracture vs Ankle Fracture-Dislocation
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 06-12-03A
Record Dates: First submitted 2013-03-28; First posted 2014-07-24 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2017-01

CONDITIONS: Ankle Fractures
Keywords: ankle fracture; ankle fracture-dislocation; prospective; observational
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ankle Fracture: Patients with isolated ankle fractures.
- Ankle Fracture-Dislocation: Patients with ankle fracture-dislocations.

SUMMARY:
The purpose of this study is to compare outcomes of patients with an ankle fracture to those with ankle fracture-dislocations. We hypothesize that long-term clinical outcomes for patients sustaining ankle fracture dislocations are poorer than those without dislocation.

DETAILED DESCRIPTION:
Orthopaedic literature has very limited data regarding outcomes following ankle fracture dislocations. Increased knowledge of the long-term consequences of these injuries could usher in changes to treatment paradigms, potentially resulting in improved outcomes. Thirty patients will be enrolled into two arms of this prospective study: isolated ankle fractures and ankle fracture dislocations. Patients will be followed through their operative and postoperative course and clinical and radiographic assessments will be analyzed. We plan to compare the clinical, radiographic, and functional outcomes of patients with ankle fractures to those with ankle fracture-dislocations. We also plan to identify factors that contribute to or predict poor clinical, functional, and/or radiographic outcomes in patients with ankle fractures and fracture-dislocations.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sustain an isolated bi-malleolar or trimalleolar ankle fracture or an ankle fracture-dislocation requiring open reduction internal fixation
* Patients ages 18 and over
* The subject is psychosocially, mentally, and physically able to understand and comply with the requirements of the study
* Open and closed fractures (excluding Gustilo grade 3)
* English must be patient's primary language

Exclusion Criteria:

* Previous injury or significant osteoarthritis to the affected ankle
* Current ipsilateral or contralateral lower extremity injury with the exception of a contralateral ankle fracture or fracture-dislocation
* Retained hardware from a previous injury at or around the tibia-talar joint of the affected extremity
* Patients under the age of 18
* History of inflammatory arthropathy
* Traumatic Brain Injury or Spinal Cord Injury preventing weightbearing on the lower extremities
* The subject has another concurrent physical or mental condition that is likely to affect compliance with the study requirements
* Patients with Gustilo grade 3B and 3C open fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be selected from Carolinas Medical Center Level I Trauma Center.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-09; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Functional Outcome | 6, 12, and 24 months
  Clinical and functional outcomes will be measured using the Foot and Ankle Ability Measure (FAAM) and the Short Form Musculoskeletal Functional Assessment (SMFA).
  Radiographic analysis will be performed to determine nonunion, malunion, joint space incongruity, hardware failure/loosening, and/or severity of osteoarthritis. The Van Dijk grading scale will be used for radiographic assessment.

SECONDARY OUTCOMES:
Radiographic Outcome | 24 month
  Radiographic analysis will be performed to determine nonunion, malunion, joint space incongruity, hardware failure/loosening, and/or severity of osteoarthritis. The Van Dijk grading scale will be used for radiographic assessment.

OTHER OUTCOMES:
Additional surgical procedures | 2 years
  Documentation of any additional surgical procedures conducted on the affected ankle. Any surgical procedure will be noted. These may include debridement for infection or dehiscence, revision for hardware failure, arthroscopy, ankle arthrodesis, or cartilage restoration procedures.
Postoperative Complications | 2 years
  Postoperative complications will be documented and analyzed to determine if there are significant differences between the two groups. These will include infection requiring antibiotics or debridement, hardware failure, nerve or vascular injury, deep venous thrombosis, or revision surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bosse, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center- Main, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data Sharing will need to be discussed with investigators.